CLINICAL TRIAL: NCT04401800
Title: A Phase 2 Study to Investigate the Preliminary Antitumor Activity, Safety and Tolerability of Tislelizumab in Combination With Lenvatinib in Patients With Unresectable Locally Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: Preliminary Antitumor Activity, Safety and Tolerability of Tislelizumab in Combination With Lenvatinib for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-211; CTR20200972 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma; Unresectable Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib With Tislelizumab (Experimental): Participants received lenvatinib based on baseline weight (12 milligrams [mg] or 8 mg once daily for participants with a baseline weight of >= 60 kilograms [kg] or < 60 kg, respectively) along with tislelizumab 200 mg on Day 1 of each 21-day cycle (once every 3 weeks) until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
  Interventions: Drug: Lenvatinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Lenvatinib — Capsules administered orally once daily
Drug: Tislelizumab — 200 mg intravenous (IV) infusion administered on Day 1 of each cycle

SUMMARY:
The primary objective of this study was to assess the preliminary antitumor activity as indicated by overall response rate (ORR) of tislelizumab in combination with lenvatinib in participants with unresectable locally advanced or metastatic hepatocellular carcinoma (HCC) by central site imaging facility per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

ELIGIBILITY:
Key Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments
2. Unresectable locally advanced or metastatic HCC, which must be confirmed by histologically or cytologically. Fibrolamellar, sarcomatoid, or mixed cholangiocarcinoma histology confirmed by histologically or cytologically is excluded.
3. Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease that is not amenable to or has progressed after loco-regional therapy and is not amenable to a curative treatment approach
4. Did not receive any systemic treatment before and is unwilling to accept standard of care treatment or not suitable for standard of care treatment as judged by investigators
5. At least 1 measurable lesion as defined by RECIST v1.1
6. European Cancer Oncology Group (ECOG) Performance Status ≤ 1
7. Child-Pugh A classification for liver function assessed within 7 days of first dose of study drugs

Key Exclusion Criteria:

1. Active autoimmune diseases or history of autoimmune diseases that may relapse
2. Any active malignancy ≤ 2 years before the first dose of study drugs except for specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)
3. Uncontrolled diabetes or > Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium despite standard medical management, or ≥ Grade 3 hypoalbuminemia ≤ 14 days before the first dose of study drugs
4. Any known brain or leptomeningeal metastases
5. Concurrent participation in another therapeutic clinical study

NOT: Other protocol defined Inclusion/Exclusion criteria may apply NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (9):
- China (9):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Xu L, Chen J, Liu C, Song X, Zhang Y, Zhao H, Yan S, Jia W, Wu Z, Guo Y, Yang J, Gong W, Ma Y, Yang X, Gao Z, Zhang N, Zheng X, Li M, Su D, Chen M. Efficacy and safety of tislelizumab plus lenvatinib as first-line treatment in patients with unresectable hepatocellular carcinoma: a multicenter, single-arm, phase 2 trial. BMC Med. 2024 Apr 23;22(1):172. doi: 10.1186/s12916-024-03356-5. PMID 38650037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 study sites in China.
Pre-assignment Details: The study consisted of two parts: Part 1 (Safety run-in part) and Part 2 (Extension part). Results were planned to be reported and analyzed combined for Part 1 (safety-run) and Part 2 of the study as all participants received the same treatment.
Period: Overall Study
Arm/Group | Lenvatinib With Tislelizumab
Started | 64
Completed | 38
Not Completed | 26
Not completed — Death | 17
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety analysis set which included all participants who received at least 1 dose of any study drug (any component for the combination therapy).
Groups:
- Lenvatinib With Tislelizumab: Participants received lenvatinib based on baseline weight (12 mg or 8 mg once daily for participants with a baseline weight of >= 60 kg or < 60 kg, respectively) along with tislelizumab 200 mg on Day 1 of each 21-day cycle (once every 3 weeks) until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 64
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Assessed by Central Imaging Facility Based on RECIST v1.1
Description: ORR was defined as the percentage of participants achieving the best overall response (BOR) of complete response (CR) or partial response (PR). The 95% confidence interval (CI) was estimated using the Clopper-Pearson method. Per Response evaluation criteria in solid tumors (RECIST) version (v)1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Response was assessed every 6 weeks for the first year and approximately every 9 weeks thereafter through December 2022; up to 27 months
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF) which included all dosed participants with measurable disease at baseline per RECIST v1.1 and who had at least one evaluable post-baseline tumor assessment unless treatment was discontinued due to clinical disease progression or death before the first post-treatment tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
percentage of participants | 38.7 [26.6 to 51.9]
Statistical Analysis 1: Comparison: Lenvatinib With Tislelizumab; Test type: Superiority; p = 0.0002, Binomial exact test

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs) and TEAEs Leading to Treatment Discontinuation and Modification
Description: A TEAE was defined as adverse event (AE) that had an onset date or a worsening in severity from baseline (pre-treatment) on or after the first dose of study drug(s) and up to 30 days following study drug(s) discontinuation or initiation of new anticancer therapy, whichever occurs first determined according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. SAE: any untoward medical occurrence at any dose: resulted in death; was life threatening; required prolong inpatient hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect or was considered a significant medical event by the investigator.
Time Frame: From the date of the first dose of study drug up to 30 days after last dose of study drug (maximum time on treatment was 12 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 64
Participants
  TEAE | 64
  TESAE | 11
  TEAE leading to treatment discontinuation | 4
  TEAE leading to dose modification | 37

3. Secondary Outcome: Objective Response Rate (ORR) as Assessed by the Investigator Based on RECIST v1.1
Description: ORR was defined as the percentage of participants achieving the BOR of CR or PR. The 95% CI was estimated using the Clopper-Pearson method. Per RECIST v1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Response was assessed every 6 weeks for the first year and approximately every 9 weeks thereafter through December 2022; i.e., up to 27 months
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
percentage of participants | 41.9 [29.5 to 55.2]
Statistical Analysis 1: Comparison: Lenvatinib With Tislelizumab; Test type: Superiority; p < 0.0001, Binomial exact test

4. Secondary Outcome: Objective Response Rate (ORR) as Assessed by the Investigator and Central Site Imaging Facility Based on Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: ORR was defined as the percentage of participants achieving the BOR of CR or PR. The 95% CI was estimated using the Clopper-Pearson method. Per modified RECIST (mRECIST), CR was defined as the disappearance of any intratumoral arterial enhancement in all target lesions. PR: at least a 30% decrease in the sum of diameters of viable (contrast enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions.
Time Frame: as for outcome 1
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
percentage of participants
  By investigator | 46.8 [34.0 to 59.9]
  By Central Site Imaging Facility | 46.8 [34.0 to 59.9]
Statistical Analysis 1: Comparison: Lenvatinib With Tislelizumab; ORR as Assessed by the Investigator; Test type: Superiority; p < 0.0001, Binomial exact test
Statistical Analysis 2: Comparison: Lenvatinib With Tislelizumab; ORR as Assessed by Central Site Imaging Facility; Test type: Superiority; p < 0.0001, Binomial exact test

5. Secondary Outcome: Objective Response Rate (ORR) as Assessed by the Investigator and Central Site Imaging Facility Based on Immune Related Response Evaluation Criteria in Solid Tumors (iRECIST)
Description: ORR was defined as the percentage of participants achieving the BOR of immune complete response (iCR) or partial response (iPR). The 95% CI was estimated using the Clopper-Pearson method. Per iRECIST, iCR was defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 mm in the short axis. iPR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. iRECIST is a modification to RECIST that considers unique patterns of atypical response in immunotherapy and enables treatment beyond initial radiographic progression.
Time Frame: as for outcome 1
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
percentage of participants
  By investigator | 43.5 [31.0 to 56.7]
  By Central Site Imaging Facility | 38.7 [26.6 to 51.9]
Statistical Analysis 1: Comparison: Lenvatinib With Tislelizumab; ORR as Assessed by the Investigator; Test type: Superiority; p < 0.0001, Binomial exact test
Statistical Analysis 2: Comparison: Lenvatinib With Tislelizumab; ORR as Assessed by Central Site Imaging Facility; Test type: Superiority; p = 0.0002, Binomial exact test

6. Secondary Outcome: Duration of Response (DOR) As Assessed by The Investigator Based on RECIST v1.1
Description: DOR was defined as the time interval between the date of the earliest qualifying response (CR or PR) and the date of PD or death (whichever occurred earlier). DOR was estimated using the Kaplan-Meier method. Per RECIST v1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From the date of earliest response to the date of first documentation of disease progression or death, whichever occurred first (up to 35 months)
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF) on the subset of participants with a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 26
months | NA [NA to NA] — Median and 95% Confidence Interval (CI) could not be calculated due to low number of participants with events.

7. Secondary Outcome: Duration of Response (DOR) As Assessed by The Central Site Imaging Facility Based on RECIST v1.1
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF) on the subset of participants with a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 24
months | NA [NA to NA] — Median and 95% CI could not be calculated due to low number of participants with events.

8. Secondary Outcome: Duration of Response (DOR) As Assessed by The Investigator Based on mRECIST
Description: DOR was defined as the time interval between the date of the earliest qualifying response (CR or PR) and the date of PD or death (whichever occurs earlier). DOR was estimated using the Kaplan-Meier method. Per mRECIST, CR was defined as the disappearance of any intratumoral arterial enhancement in all target lesions. PR: at least a 30% decrease in the sum of diameters of viable (contrast enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions. PD: an increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since the treatment started.
Time Frame: as for outcome 6
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF) on the subset of participants with a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 29
months | 9.7 [5.6 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with events.

9. Secondary Outcome: Duration of Response (DOR) As Assessed by the Central Site Imaging Facility Based on mRECIST
Description: as for outcome 8
Time Frame: as for outcome 6
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF) on the subset of participants with a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 29
months | NA [NA to NA] — Median and 95% CI could not be calculated due to low number of participants with events.

10. Secondary Outcome: Duration of Response (DOR) As Assessed by The Investigator Based on iRECIST
Description: DOR was defined as the time interval between the date of the earliest qualifying response (iCR or iPR) and the date of confirmed progressive disease (iCPD) or death (whichever occurs earlier). DOR was estimated using the Kaplan-Meier method. Per iRECIST, iCR was defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 mm in the short axis. iPR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. iRECIST is a modification to RECIST that considers unique patterns of atypical response in immunotherapy and enables treatment beyond initial radiographic progression.
Time Frame: as for outcome 6
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF) on the subset of participants with a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 27
months | NA [9.7 to NA] — Median and Upper limit of 95% CI could not be calculated due to low number of participants with events.

11. Secondary Outcome: Duration of Response (DOR) As Assessed by The Central Site Imaging Facility Based on iRECIST
Description: as for outcome 10
Time Frame: From the date of earliest response to the date of first documentation of disease progression or death, whichever occurs first (up to 35 months)
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF) on the subset of participants with a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 24
months | NA [NA to NA] — Median and 95% CI could not be calculated due to low number of participants with events.

12. Secondary Outcome: Disease Control Rate (DCR) As Assessed by The Investigator and Central Site Imaging Facility Based on RECIST v1.1
Description: DCR was defined as the percentage of participants with BOR of CR, PR or SD. Participants without post-baseline tumor assessment were considered as failure in DCR. The 95% CI was estimated using the Clopper-Pearson method. Per RECIST v1.1., CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 1
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
percentage of participants
  By investigator | 85.5 [74.2 to 93.1]
  By Central Site Imaging Facility | 90.3 [80.1 to 96.4]

13. Secondary Outcome: Disease Control Rate (DCR) As Assessed by The Investigator and Central Site Imaging Facility Based on mRECIST
Description: DCR was defined as the percentage of participants with BOR of CR, PR or SD. Participants without post-baseline tumor assessment were considered as failure in DCR. The 95% CI was estimated using the Clopper-Pearson method. Per mRECIST, CR was defined as the disappearance of any intratumoral arterial enhancement in all target lesions. PR: at least a 30% decrease in the sum of diameters of viable (contrast enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions. Stable disease (SD): any cases that do not qualify for either partial response or progressive disease.
Time Frame: as for outcome 1
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
percentage of participants
  By investigator | 85.5 [74.2 to 93.1]
  By Central Site Imaging Facility | 90.3 [80.1 to 96.4]

14. Secondary Outcome: Disease Control Rate (DCR) As Assessed by The Investigator and Central Site Imaging Facility Based on iRECIST
Description: DCR was defined as the percentage of participants with BOR of iCR, iPR or immune stable disease (iSD). Participants without post-baseline tumor assessment were considered a failure in DCR. The 95% CI was estimated using the Clopper-Pearson method. Per iRECIST, iCR was defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 mm in the short axis. iPR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. iSD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. iRECIST is a modification to RECIST that considers unique patterns of atypical response in immunotherapy and enables treatment beyond initial radiographic progression.
Time Frame: as for outcome 1
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
percentage of participants
  By investigator | 88.7 [78.1 to 95.3]
  By Central Site Imaging Facility | 90.3 [80.1 to 96.4]

15. Secondary Outcome: Progression Free Survival (PFS) As Assessed by The Investigator Based on RECIST v1.1
Description: PFS was defined as the time from the date of the first dose of study drug(s) to the date of the confirmed documentation of PD or death, whichever occurred first. PFS was estimated using the Kaplan-Meier method. Per RECIST v1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From date of first dose of study drug until the date of first documented progression or date of death from any cause, whichever came first (up to 35 months)
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
months | 9.6 [5.3 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with PFS events.

16. Secondary Outcome: Progression Free Survival (PFS) As Assessed by The Central Site Imaging Facility Based on RECIST v1.1
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
months | 8.2 [6.8 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with PFS events.

17. Secondary Outcome: Progression Free Survival (PFS) As Assessed by The Investigator Based on mRECIST
Description: PFS was defined as the time from the date of the first dose of study drug(s) to the date of the confirmed documentation of PD or death, whichever occurs first. PFS was estimated using the Kaplan-Meier method. Per mRECIST, PD was defined as an increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since the treatment started.
Time Frame: as for outcome 15
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
months | 6.9 [4.2 to 9.6]

18. Secondary Outcome: Progression Free Survival (PFS) As Assessed by The Central Site Imaging Facility Based on mRECIST
Description: as for outcome 17
Time Frame: as for outcome 15
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
months | 8.3 [6.7 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with PFS events.

19. Secondary Outcome: Progression Free Survival (PFS) As Assessed by The Investigator Based on iRECIST
Description: PFS was defined as the time from the date of the first dose of study drug(s) to the date of the confirmed documentation of progressive disease (iCPD) or death, whichever occurs first. PFS was estimated using the Kaplan-Meier method. Per iRECIST v1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. iRECIST is a modification to RECIST that considers unique patterns of atypical response in immunotherapy and enables treatment beyond initial radiographic progression.
Time Frame: as for outcome 15
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
months | 11.1 [6.8 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with PFS events.

20. Secondary Outcome: Progression Free Survival (PFS) As Assessed by The Central Site Imaging Facility Based on iRECIST
Description: as for outcome 19
Time Frame: as for outcome 15
Population: Analysis was performed on Efficacy-Evaluable Analysis Set (EFF).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib With Tislelizumab
Number analyzed (Participants) | 62
months | 8.2 [6.8 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with PFS events.

ADVERSE EVENTS:
Time Frame: All-cause mortality data were collected through the end of the study, up to 35 months. Adverse events were collected from first dose up to 30 days after last dose; maximum time on treatment was 12 months
Description: Analysis was performed on safety analysis set.
Groups:
- Tislelizumab + Lenvatinib: Participants received lenvatinib based on baseline weight (12 mg or 8 mg once daily for participants with a baseline weight of >= 60 kg or < 60 kg, respectively) along with tislelizumab 200 mg on Day 1 of each 21-day cycle (once every 3 weeks) until disease progression, unacceptable toxicity, or withdrawal for other reasons, whichever occurred first.
Arm/Group | Tislelizumab + Lenvatinib
All-Cause Mortality (participants affected / at risk) | 17/64
Serious Adverse Events (participants affected / at risk) | 11/64
Other Adverse Events (participants affected / at risk) | 63/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Lenvatinib (N=64)
Retinal detachment (Eye disorders) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Death (General disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Lenvatinib (N=64)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 3 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4)
Sinus bradycardia (Cardiac disorders) | 3 (5)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 20 (20)
Thyroid disorder (Endocrine disorders) | 4 (4)
Thyroid mass (Endocrine disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 11 (18)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gingival swelling (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 4 (4)
Toothache (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 6 (8)
Pyrexia (General disorders) | 4 (7)
Hepatic function abnormal (Hepatobiliary disorders) | 5 (7)
Pharyngitis (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 5 (5)
Alanine aminotransferase increased (Investigations) | 8 (9)
Amylase increased (Investigations) | 11 (15)
Aspartate aminotransferase increased (Investigations) | 22 (25)
Bilirubin conjugated increased (Investigations) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 8 (9)
Blood bilirubin increased (Investigations) | 12 (20)
Blood chloride decreased (Investigations) | 3 (3)
Blood creatine phosphokinase MB increased (Investigations) | 10 (20)
Blood creatine phosphokinase increased (Investigations) | 8 (12)
Blood creatinine increased (Investigations) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 11 (14)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2)
C-reactive protein increased (Investigations) | 5 (11)
Electrocardiogram ST segment abnormal (Investigations) | 2 (2)
Electrocardiogram ST-T change (Investigations) | 3 (3)
Electrocardiogram T wave abnormal (Investigations) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 7 (7)
Glomerular filtration rate decreased (Investigations) | 2 (2)
Lipase increased (Investigations) | 12 (14)
Lymphocyte count decreased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 6 (11)
Platelet count decreased (Investigations) | 17 (28)
Prealbumin decreased (Investigations) | 2 (2)
Thyroid function test abnormal (Investigations) | 3 (4)
Total bile acids increased (Investigations) | 4 (8)
Urinary occult blood positive (Investigations) | 2 (2)
Weight decreased (Investigations) | 20 (24)
White blood cell count decreased (Investigations) | 8 (14)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 7 (15)
Proteinuria (Renal and urinary disorders) | 29 (60)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 8 (9)
Hypertension (Vascular disorders) | 23 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-12-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT04401800/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT04401800/SAP_001.pdf